CLINICAL TRIAL: NCT03058731
Title: Comparison of Symptomatic and Radiographic Outcomes of Paraesophageal Hernia Repair With and Without MatriStem Surgical Matrix
Brief Title: ACELL Mesh for Paraesophageal Hernia Repair
Status: Completed | Type: Observational
Sponsor: University of South Florida (Other)
Collaborators: Integra LifeSciences Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: ACELL01
Record Dates: First submitted 2017-02-16; First posted 2017-02-23 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Paraesophageal Hernia
MeSH Terms: conditions — Hernia, Hiatal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Matristem: Hernia repair with MatriStem Surgical Matrix
  Interventions: Device: Matristem
- Control: Other biological mesh
  Interventions: Device: Control

INTERVENTIONS:
Device: Matristem — Paraesophageal hernia repair with MatriStem Surgical Matrix
  Groups: Matristem
Device: Control — Paraesophageal hernia repair with other biologic mesh
  Groups: Control

SUMMARY:
This is a prospective, case-matched, systematic follow up of up to 70 pre-existing patients whom underwent paraesophageal hernia repair between June 1, 2012 and September 30, 2016. Patients whom are willing to participate in the study will be asked to return for a one time follow up visit to reassess for hiatal hernia recurrence both symptomatically and radiologically to compare the efficacy of the use of MatriStem Surgical Matrix (ACell) mesh to other biologic meshes.

DETAILED DESCRIPTION:
The participating "MatriStem" patients (N=35) will be matched to "control" patients who were treated surgically by Dr. Vic Velanovich or Dr. Michael Albrink for paraesophageal hernia with a biological mesh other than MatriStem Surgical Matrix (N=35) during the study timeframe at Tampa General Hospital. Patients will be matched by age (+ 5 years), gender, and operative approach (laparoscopic, laparotomy, or thoracic approach).

Study participation will require only one visit. Once the patient signs the consent form, operative details and the postoperative course will be reviewed retrospectively.

Visit 1 (≥ 12 months post-PEHR)

1. Review the study with the subject and/or subject's legal representative, and obtain written informed consent and HIPAA authorization.
2. Assign the subject a unique screening/enrollment number (assigned sequentially starting from 001).
3. Pregnancy test if subject is of childbearing potential
4. Confirm subject eligibility.
5. Record demographics data, which includes date of birth, race, ethnicity, and gender.
6. Record current clinical symptoms in relation to the HH.
7. Record medications, including over-the-counter and herbal medications, taken postoperatively in relation to the HH.
8. Record medical history with respect to the paraesophageal hernia prior to the surgical repair. If available, the following information will be recorded: hernia type, hernia size, organo-axial, or meso-axial rotation, and operative approach (laparoscopic, laparotomy, or thoracic approach).
9. Record medical history with respect to the paraesophageal hernia after the surgical repair (size of mesh implant, length of surgery [calculated as the time from incision to wound closure], postoperative complications to include need for reoperation, mesh migration, reherniation, etc [from date of hospital discharge to study visit], and symptom frequency).
10. Perform esophagogram at TGH.
11. Administer GERD-HRQL symptom severity questionnaire.
12. Administer SF-36 generic quality of life instrument.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Underwent primary or re-do PEHR with biological mesh by Dr. Vic Velanovich or Dr. Michael Albrink between June 1, 2012 and September 30, 2016
* Written informed consent obtained from subject prior to esophagogram procedure and ability for subject to comply with the requirements of the study

Exclusion Criteria:

* Age < 18 years of age
* Underwent PEHR by a surgeon other than Dr. Vic Velanovich or Dr. Michael Albrink
* Underwent PEHR outside of the timeframe of June 1, 2012 and September 30, 2016
* Subject is involved in ongoing medical litigation, confirmed via subject report
* Subject is incarcerated, confirmed via subject report
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients that had a PEHR performed with a biological mesh between June 1, 2012 and September 30, 2016 at Tampa General Hospital
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2016-02-02 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2019-01-28 (Actual)

PRIMARY OUTCOMES:
Rate of hernia recurrence | 12 months

SECONDARY OUTCOMES:
Mean vertical height of hiatal hernia | 12 months
  For patients with hiatal hernia recurrence
Mean cross-sectional area of hiatal hernia | 12 months
  For patients with hiatal hernia recurrence
Rate of postoperative complications | 12 months
Mean GERD-Health Related QOL score | 12 months
Mean SF-36 QOL score | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Vic Velanovich, MD, Principal Investigator — University of South Florida
Locations (1):
- Tampa General Hospital, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oelschlager BK, Pellegrini CA, Hunter JG, Brunt ML, Soper NJ, Sheppard BC, Polissar NL, Neradilek MB, Mitsumori LM, Rohrmann CA, Swanstrom LL. Biologic prosthesis to prevent recurrence after laparoscopic paraesophageal hernia repair: long-term follow-up from a multicenter, prospective, randomized trial. J Am Coll Surg. 2011 Oct;213(4):461-8. doi: 10.1016/j.jamcollsurg.2011.05.017. Epub 2011 Jun 29. PMID 21715189
- [Background] Oelschlager BK, Pellegrini CA, Hunter J, Soper N, Brunt M, Sheppard B, Jobe B, Polissar N, Mitsumori L, Nelson J, Swanstrom L. Biologic prosthesis reduces recurrence after laparoscopic paraesophageal hernia repair: a multicenter, prospective, randomized trial. Ann Surg. 2006 Oct;244(4):481-90. doi: 10.1097/01.sla.0000237759.42831.03. PMID 16998356
- [Result] Hashemi M, Peters JH, DeMeester TR, Huprich JE, Quek M, Hagen JA, Crookes PF, Theisen J, DeMeester SR, Sillin LF, Bremner CG. Laparoscopic repair of large type III hiatal hernia: objective followup reveals high recurrence rate. J Am Coll Surg. 2000 May;190(5):553-60; discussion 560-1. doi: 10.1016/s1072-7515(00)00260-x. PMID 10801022
- [Result] Mattar SG, Bowers SP, Galloway KD, Hunter JG, Smith CD. Long-term outcome of laparoscopic repair of paraesophageal hernia. Surg Endosc. 2002 May;16(5):745-9. doi: 10.1007/s00464-001-8194-7. Epub 2002 Feb 8. PMID 11997814